CLINICAL TRIAL: NCT02780635
Title: Use of Mobile Apps for Those With PTSD and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Owen, Clinical Psychologist, VA Palo Alto Health Care System
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 33003
Record Dates: First submitted 2016-05-04; First posted 2016-05-23 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Ptsd
Keywords: family, caregiving, ptsd, couples
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- App + Couples Coach Intervention (Experimental): Both members of the couple will receive a mobile app for PTSD: PTSD Coach for the Veteran and PTSD Family Coach for the partner/spouse. Those assigned to this arm will also receive mailed materials that are designed to help increase positive communication strategies.
  Interventions: Behavioral: Mobile App + Mailed Materials for managing stress associated with PTSD; Behavioral: Mobile App for managing stress associated with PTSD
- App Alone (Active Comparator): Both members of the couple will receive a mobile app for PTSD: PTSD Coach for the Veteran and PTSD Family Coach for the partner/spouse.
  Interventions: Behavioral: Mobile App for managing stress associated with PTSD

INTERVENTIONS:
Behavioral: Mobile App + Mailed Materials for managing stress associated with PTSD — PTSD Coach and PTSD Family Coach mobile apps plus mailed "Couples Coach" intervention materials and discussion board added to PTSD Family Coach app
  Arms: App + Couples Coach Intervention
Behavioral: Mobile App for managing stress associated with PTSD — PTSD Coach and PTSD Family Coach mobile apps

SUMMARY:
In layperson's language state the purpose of the study in 3-5 sentences.

Previous research has demonstrated that intimate partners can positively influence those with PTSD to seek treatment. The investigators have preliminary evidence to demonstrate that mobile apps, such as PTSD Coach can be helpful for those with PTSD, and the current study will provide Veterans with PTSD and their partners with a mobile app designed to promote engagement with evidence-based treatments for PTSD. The purpose of this PILOT study is to evaluate methods for delivering a couples-based intervention to reduce PTSD symptoms and improve relationship quality in Veterans and their intimate partners.

b) State what the Investigator(s) hope to learn from the study. Include an assessment of the importance of this new knowledge.

Understanding ways to improve the public health impact of public-facing, evidence-based mobile apps is critical. This study will test a low-cost, "high-touch" approach to improving the outcomes associated with use of the PTSD Coach and PTSD Family Coach mobile apps,which are already available to the general public and used by over 55,000 new users per year.This study will test whether the involvement of an intimate partner in the use of a mobile app for PTSD will result in changes in how the mobile apps are used and in relationship quality and PTSD symptoms over time. Additionally, this study will test whether the addition of a discussion board can improve engagement with the apps and/or outcomes. The study will also provide useful qualitative data that can inform the development of subsequent dyadic interventions using mobile technologies.

c) Explain why human subjects must be used for this project. (i.e. purpose of study is to test efficacy of investigational device in individuals with specific condition; purpose of study is to examine specific behavioral traits in humans in classroom or other environment)

The purpose of this study is to evaluate how Veterans and their partners interact with evidence-based mobile apps for improving PTSD symptoms.

DETAILED DESCRIPTION:
Please SUMMARIZE the research procedures, screening through closeout, which the human subject will undergo. Refer to sections in the protocol attached in section 16, BUT do not copy the clinical protocol. Be clear on what is to be done for research and what is part of standard of care.

In brief, the study team will attempt to recruit 100 couples in which one partner is a community-dwelling Veteran with significant, untreated symptoms of posttraumatic stress disorder (PTSD) symptoms. All participants will receive access to a mobile app designed by Veterans Affairs (VA). Veterans will receive access to the PTSD Coach mobile app, and their partners will receive access to the PTSD Family Coach mobile app. Potential participants will be identified from targeted Facebook and other social media outreach efforts. Those who view an advertisement will be directed to the study website, hosted by Stanford's Qualtrics domain, where they will be provided with information about the study, screened for eligibility,and then provided with an informed consent document. Upon completing the informed consent process, participants will be asked to complete a baseline survey and then to share information about the study with their partner. Veterans and their partners will be connected only by a subject identification number. After completing the baseline survey, all participants will then be encouraged to use the PTSD Coach app or the PTSD Family Coach app as often or as little as they like.

Using random assignment, half of the dyads will also be provided with a) access to a secure, confidential discussion board, where they will be able to post new messages and respond to messages posted by others and b) mailed information packages that contain information about coping with PTSD, coping with a spouse's PTSD, and strategies for managing relationship distress associated with PTSD. Those dyads who do not receive access to the discussion board will still receive access to the mobile apps but will not have access to either the discussion board or the mailed information packages.

Outcomes will be evaluated using objective measures of engagement with the apps, changes in attitudes toward use of mental health services, relationship quality,changes over time in PTSD and stress symptoms, and qualitative experiences associated with use of the apps. Barriers to implementation and identified strategies for overcoming barriers will be catalogued over the duration of the study.

Description of PTSD Coach:

Participants will be provided with a link to download PTSD Coach (freely available on iTunes and Google Play Stores or through myvaapps.com) and brief recommendations for how to use the app over the subsequent 8 weeks of the study. PTSD Coach is a mobile app for iPhone and Android, developed by the VA National Center for PTSD in collaboration with National Center for Telehealth and Technology (T2) and the Department of Veterans Affairs Patient Care Services. PTSD Coach was initially developed and launched in March, 2011, with usability and focus group data derived from a sample of 80 veterans with PTSD, many of whom were explicitly requesting "something I can do when I'm stressed, wherever I am." The app provides 4 primary treatment components: 1) psychoeducation about PTSD, 2) self-monitoring tools, 3) immediate tools for symptom management, and 4) immediate access to public and private support resources. The psychoeducation component provides text and audio informational topics about PTSD, with an emphasis on normalizing the condition, and information about ways to begin engaging with mental health services. The self-monitoring tools component administers the PTSD Checklist Civilian version (PCL-C), provides tailored feedback on symptom level and changes since the last assessment, and allows and encourages users to create reminders to self-monitor their symptom levels. The symptom management component provides specific tools tailored for managing reminders of trauma, avoiding trauma-related triggers, overcoming feelings of being disconnected from others, overcoming feelings of being disconnected from reality,improving sleep, and reducing feelings of sadness, hopelessness, worry, anxiety, or anger.These tools include audio-based relaxation exercises, guided deep breathing, making plans for social activities, engaging in pleasant activities, tips for distraction from unpleasant sensations, and other simple exercises. The support component encourages users to create a personal support network (from their phone's contact list) and provides users with information about additional resources for veterans (e.g., crisis and help-line numbers). Evidence for PTSD Coach is described in detail in the Preliminary Studies section. In brief, use of PTSD Coach alone is associated with significant within-session changes in ratings ofdistress43 and demonstrates a small but clinically meaningful effect on PTSD symptoms(d=.30, f~.15) relative to a wait-list control group.

Partners will be provided with a link to the PTSD Family Coach app. PTSD Family Coach provides four main intervention elements: Learn, Support, Tools for Managing Stress, and Self-Assessment. The "Learn" section of the app provides extensive, mobile-friendly information about the basics of PTSD and how to best support their loved one with PTSD, how to take care of on self while living with someone with PTSD, how to take care of relationships with children and with one's partner, and how to most effectively encourage their partner to engage in professional care. The "Support" section of the app provides information about how to get immediate crisis help (e.g., for medical emergencies, suicidal thoughts, or threats of violence), how to get help in talking with a partner about PTSD, how to find family-specific services, resources for parents and children, and resources for the Veteran. The "Tools for Managing Stress" section of the app contains interactive relaxation tools, cognitive strategies for managing stress, mindfulness exercises, encouragement to engage in pleasant activities and to engage in social activities, safety-planning tools, tips for good sleep hygiene, and grounding techniques. Finally, the "Self-Assessment" section of the app provides tools for self-monitoring stress symptoms and tracking these symptoms over time.Description of the Discussion Boards to be used in this study:All discussion boards will be privately hosted on the secure https://www.health-space.net sight maintained by the PI and can only be accessed with a unique API key and valid invitation code stored in the mobile app, so that only those who have been provided with both a research version of the study app and a valid invitation code will be able to access the discussion board. There will be 2 unique discussion boards: one for family members (i.e., accessed from the PTSD Family Coach app) and one for Veterans (i.e., accessed from the PTSD Coach app). Those who choose to post a message to the discussion board will be identified only by their invitation code (a random string of 6 characters and/or digits), and all messages will be reviewed by the investigators in order to ensure safety and appropriateness before they can be viewed by any other participants. As soon as a message is posted, an automated email will be sent to each of the investigators, who will be asked to log-in to a secure website in order to approve the submitted message so that it can viewed by other participants. Should any safety or privacy-related concerns arise, or the message is deemed inappropriate for any other reason, the participant who submitted the message will be contacted and provided with additional information necessary for either obtaining additional assistance or modifying the message to make more appropriate or private as necessary.

Every 2 weeks for 8 weeks, each participant will be mailed an information packet (i.e., 4 packets in total for each participant) that will provide additional information on managing stress and conflict in relationships,increasing positive interactions in the relationship, problem-solving in relationships, and increasing positive communication in relationships. Information packets will contain general information, a list of available resources that can provide additional information, and suggested exercises to practice with their partner or by using the mobile app.

Ten weeks after being randomized, Veterans and their partners will be asked to complete a follow-up survey using the Qualtrics web survey tool. Those participants who are willing to take part in a telephone interview will be contacted by telephone to participate in a 30-minute qualitative interview about the app, communication with their partner about PTSD symptoms,and suggestions for optimizing partner-based interventions using mobile apps.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate, participants must be either a Veteran with PTSD or living with a partner who is a Veteran with PTSD.

Veterans must be:

1. A veteran of the U.S. Armed Forces
2. Must have a previous diagnosis of PTSD
3. Must have access to a smart phone using the iOS operating system
4. Must not have previously used PTSD Coach.

Partners of Veterans must be:

1. An intimate partner of a Veteran
2. Living with that partner
3. Must have access to a smart phone using the iOS operating system
4. must be experiencing significant stress

Exclusion Criteria:

a) actual or threatened interpersonal violence in the home

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden | 10 weeks
  Montgomery Burden Interview
Functional Well-Being | 10 weeks
  Partner-rated Interpersonal Well-Being Scale
Personal Health Questionnaire Depression Scale | 10 weeks
  8 Item scale measuring depression.
Generalized Anxiety Symptoms | 10 weeks
  Generalized Anxiety Disorder-7 Scale (GAD-7)
PTSD Symptoms | 10 weeks
  5 Item Partner-rated Posttraumatic Stress Disorder Checklist-5 (PCL-5)
Positive Relationship Behaviors | 10 weeks
  Author-constructed relationship behaviors scale
Stress | 10 weeks
  Perceived Stress Scale

SECONDARY OUTCOMES:
Emotional Intimacy | 10 weeks
  Personal Assessment of Intimacy in Relationships (PAIR) Scale
Caregiving Self-Efficacy Scale | 10 weeks
  Author-constructed questionnaire
Positive Partner Communication | 10 weeks
  Measured with items combined from the Social Constraints Scale and Communication Danger Signs Scale
Relationship Self-Efficacy | 10 weeks
  Author-constructed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System Menlo Park Division, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Undecided